CLINICAL TRIAL: NCT02960542
Title: Healthy Living Partnerships to Prevent Cancer (HELP PC) Pilot Study
Brief Title: HELP Prevent Cancer Pilot Study
Acronym: HELP PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); Danville Regional Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00039102
Record Dates: First submitted 2016-10-31; First posted 2016-11-09 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Cancer
Keywords: lifestyle intervention; weight-loss
MeSH Terms: conditions — Obesity; Neoplasms; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Weight Loss (Experimental): The Behavioral: HELP Prevent Cancer Intervention is a lifestyle intervention consisting of 24-weekly group meetings led by a community health worker and 3 individual sessions with a nutritionist/diabetes educator
  Interventions: Behavioral: HELP Prevent Cancer Intervention

INTERVENTIONS:
Behavioral: HELP Prevent Cancer Intervention — This Behavioral: Lifestyle Weigh Loss Intervention involves a dietary weight-loss program and an increase in caloric expenditure through moderate physical activity. The primary treatment objectives for the weight-loss component of the intervention will be to decrease caloric intake in a nutritionally sound manner so as to produce a weight-loss of .3 kg/week for a total weight loss of 5-7%. The primary objective for the physical activity component of the intervention will be to promote an increase in home-based energy expenditure to an eventual goal of 180 minutes/week.

SUMMARY:
This pilot study is designed to adapt a community-based diabetes prevention program to reach adults at risk for cancer.

DETAILED DESCRIPTION:
The Healthy Living Partnerships to Prevent Diabetes (HELP PD) study successfully translated the Diabetes Prevention Program (DPP) weight-loss lifestyle intervention in Winston-Salem, North Carolina by delivering the intervention via a partnership between a local diabetes education program with lay community health workers. This study documented a 7% weight loss and 4 mg/dl decrease in fasting blood glucose in patients with prediabetes in 1 year at promote healthy weight loss (1-2 pounds per week). These lifestyle strategies significantly lower costs than the DPP. The HELP PD lifestyle intervention focuses on restricting calories (while improving dietary quality) and increasing physical activity to allow participants to achieve an energy deficient state to are essential to reduce risk for type 2 diabetes but also for a multitude of chronic diseases where excess body weight plays a critical role in the development and exacerbation of the disease. In light of the community-based partnership on which HELP PD was based and the relatively low costs of program administration, the HELP PD model has the potential to be a highly effective and sustainable long-term approach to cancer prevention as well. This pilot study will be the initial step to determine feasibility of implementing the Healthy Living Partnerships to Prevent Cancer (HELP PC) in the Dan River Region of Southern Virginia through a partnership between researchers and colleagues from Wake Forest Comprehensive Cancer Center, Virginia Polytechnic Institute and State University, Danville Hematology and Oncology at the Danville Regional Medical Center, Resource Center of Southern Virginia in Danville, and Danville Regional Medical Center. Wake Forest will serve as the lead site in this study.

ELIGIBILITY:
Inclusion Criteria:

* English Proficiency: Able to read/understand English at or above a level sufficient to comprehend recruitment and intervention materials.
* Body Mass Index: BMI > 25 kg/m2.

Exclusion Criteria:

* Weight Loss: Currently involved in a supervised program for weight loss.
* Medications: Use of insulin or other diabetes medications that would require additional medical monitoring during weight-loss; use of medications for weight loss or that may impact weight or glucometabolic function (e.g. corticosteroids).
* Recent History of Cardiovascular Disease: Clinical history of cardiovascular disease (CVD) occurring within the past 6 months, including myocardial infarction, angina, coronary revascularization, stroke, transient ischemic attack (TIA), carotid revascularization, peripheral arterial disease, and congestive heart failure.
* Hypertension: Uncontrolled high blood pressure: BP > 160/100. Persons can be re-screened after controlled.
* Pregnancy: Pregnancy, breast feeding, or planning pregnancy within 1 year.
* Other Chronic Conditions: Other chronic disease likely to limit lifespan to less than 2-3 years, including any cancer requiring treatment in past 5 years except non-melanoma skin cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Recruitment of 20 eligible study participants | 6 months
  Develop and evaluate a feasible referral system to facilitate participant enrollment into the HELP PC intervention (measured by number screened and enrolled)
Retention of study participants | 6 months
  Measure retention to the HELP PC intervention (measured by number of participants attending the closeout visit after 26 weeks of intervention)
Attendance at group sessions | 6 months
  Assess participant adherence to attending the HELP PC intervention sessions (measured by community health worker documentation of session attendance)

SECONDARY OUTCOMES:
Blood Pressure | 6 months
  Estimate the means and standard deviations at baseline and 6 months.
Weight | 6 months
  Estimate the means and standard deviations at baseline and 6 months.
Glucose | 6 months
  Estimate the means and standard deviations at baseline and 6 months.
Insulin | 6 months
  Estimate the means and standard deviations at baseline and 6 months.
Cholesterol | 6 months
  Estimate the means and standard deviations at baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Z Vitolins, DrPH MPH RDN, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Danville Regional Medical Center, Danville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wise Thomas S, Blackwell Young C, Zoellner J, Brock DP, Isom S, Vitolins M. Feasibility of an Adapted Community-Based Lifestyle Intervention to Prevent Cancer in the Rural South: Healthy Living Partnerships to Prevent Cancer (HELP PC). J Cancer Educ. 2023 Apr;38(2):440-447. doi: 10.1007/s13187-022-02137-z. Epub 2022 Jan 25. PMID 35076863